CLINICAL TRIAL: NCT03633240
Title: Emergency Room Visits and Older Patients: Assessment of Jewish General Hospital Program Screening Frail Users
Brief Title: Emergency Room Visits and Older Patients (ER2)
Acronym: ER2
Status: Completed | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: CODIM-16 315
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Emergencies; Length of Stay
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ER assessment — To measure the effects of recommendations of ER2, the investigators will use ER users who will have an ER2 assessment without any recommendations as the referent group the older. This choice is possible because ER2 will be integrated into ER care in two steps:
  The first step will be limited to its assessment component in order to learn how to use the tool.
  The second step will be to follow the recommendations provided after the assessment.
  Participants will follow-up during their hospitalization via a review of their chart. They will be censored when they will be discharged from the JGH or when the duration of hospitalization will exceed 31 days.

SUMMARY:
Today's population is living longer than prior generations. Senior patients, defined as 65 years or older, are therefore increasing in number, and representing a larger number of hospitalized patients. Thus, assessing and addressing the needs of the growing number of older ER users is essential. The overall objective of the study is to examine the feasibility and the epidemiology of two screening tools ("Programme de Recherche sur l'Intégration des Services pour le Maintien de l'Autonomie" (PRISMA-7) and Emergency Room Evaluation and recommendations (ER2)) used in the Emergency Room of Jewish General Hospital to screen older patients (i.e.; ≥65 years) at risk of adverse health events. A prospective observational cohort design will be used for the study's two phases; phase 1- assessment and phase 2- assessment as well as recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Unplanned ER visits.

Exclusion Criteria:

* Death within the 24 hours of first visiting ER.
* Palliative care due to ER visit.

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: They will be separated in four main groups:
  1. Those without any PRISMA-7 and ER2.
  2. Those with PRISMA-7 and without ER2.
  3. Those with ER2 and without PRISMA-7.
  4. Those with PRISMA-7 and ER2. Each group of participants with PRISMA-7 and ER2 will be divided in two subgroups: those with all items completed and a score, and those with incomplete tools.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of using both tools in the ER | 1 day
  Percentage of participants with complete filed tools (older patients with tools filed / (older patients visiting the ER) x 100) will be calculated.
Prevalence of tools filed | 1 day
  Prevalence will be calculated for PRISMA-7, ER2 and pooled tools respectively.

SECONDARY OUTCOMES:
Feasibility of tools | 1 day
  Estimation of quality of filling using the percentage of items filled in for participants with an incomplete tool.
Length of stay | 1 day
  The LHS will be calculated using the administrative registry of the JGH and will correspond to the delay in days between the first day of admission to ED and the last day of hospitalization in the acute ward(s).
Acute medical events | 1 day
  Acute medical events occurring during the period of the ER visit and admission to the medical or surgery ward (acute organ failure, nosocomial infection, fall or death)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, Principal Investigator — Jewish General Hospital - Lady Davis Institute
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beauchet O, Afilalo M, Allali G, Lubov J, Galery K, Launay CP. "Emergency Room Evaluation and Recommendations" and Incident Hospital Admissions in Older People with Major Neurocognitive Disorders Visiting Emergency Department: Results of an Experimental Study. Dement Geriatr Cogn Disord. 2022;51(3):291-296. doi: 10.1159/000524533. Epub 2022 May 12. PMID 35551122